CLINICAL TRIAL: NCT02818088
Title: Cognitive Training in Patients With Obsessive Compulsive Disorder
Brief Title: Cognitive Training in Obsessive Compulsive Disorder
Acronym: CTOCD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The app platform was cancelled and key personnel withdrew from the project
Sponsor: University of Stellenbosch (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Principal Investigator, Christine Lochner, Professor Christine Lochner, University of Stellenbosch
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S14/05/113
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Training

ARMS (1):
- Cognitive Training (Experimental): Cognitive Training - n Back.
  Interventions: Behavioral: n-Back (Cognitive Training)

INTERVENTIONS:
Behavioral: n-Back (Cognitive Training)

SUMMARY:
This unique study will allow us to observe the neural correlates associated with working memory in an obsessive compulsive disorder (OCD) paradigm. We believe that developing working memory in participants suffering with OCD will reduce the severity of their symptomology. This will allow a greater understanding into the functioning of these participants which in turn presents with treatment possibilities.

DETAILED DESCRIPTION:
It is currently unclear whether cognitive training using a working memory task, is effective in reducing obsessive-compulsive symptoms and neuropsychological deficits in patients with OCD. Two groups (OCD and control) will be recruited. Both groups will undergo an intervention consisting of 8 weeks of cognitive training. Working memory, neuropsychological functioning and OCD symptomatology will be assessed pre and post-treatment, in both groups. Furthermore neuroimaging using functional magnetic resonance imaging (fMRI) will be conducted at baseline as well as at the end of the 8 week period in both groups. The scan will serve to show any structural or functional changes in the frontostriatal area involved with working memory. To our knowledge, this is one of the first studies to date to examine whether cognitive training improves symptoms in OCD.

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of OCD, with a score > 16 on the Yale-Brown Obsessive Compulsive Scale (YBOCS) (Goodman et al, 1989b, 1006-1011).
* Participants must be aged older than 18 and younger than 65 years.
* Right handed.
* If taking SSRI's the participant needs to be on a stable dose for at least 2 months.

Exclusion Criteria:

* Significant physical or neurological illnesses. An exception will be made for patients taking SSRI's (and not using any other drugs).
* Any significant current DSM disorder (in addition to OCD).
* Past history of significant substance or alcohol abuse.
* Pregnancy.
* Any metal pins/ prostheses or cardiac pacemakers.
* Sufferers of claustrophobia.
* Head injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-02; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (YBOCS) | Immediately after intervention
Cambridge neuropsychological test automated battery (CANTAB) | Immediately after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Stellenbosch University, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No